CLINICAL TRIAL: NCT02798419
Title: Active-Controlled Study to Assess the Efficacy and Safety of DFD-05 in Subjects With Common Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddys Laboratories, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFD05-CD-001
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Common Warts
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFD05 Cream (Experimental): DFD05 Cream
  Interventions: Drug: DFD05 Cream
- Active01 Cream (Active Comparator): Active01 Cream
  Interventions: Drug: Active01 Cream

INTERVENTIONS:
Drug: DFD05 Cream
  Arms: DFD05 Cream
Drug: Active01 Cream
  Arms: Active01 Cream

SUMMARY:
DFD05 vs. Active01 in the treatment of common warts

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, any gender or race, must be in good general health as determined by the Investigator with a clinical diagnosis of common warts.
2. Subjects must have at least 1 visible, discrete, common wart with at least a 3 mm longitudinal diameter on the hands, feet (excluding soles) and palms (in that order of priority).
3. The warts must have been present for at least the past 12 weeks, but not more than 3 years
4. Subjects must agree to only use the study products and to not use any other wart-removing product (prescription, OTC or occlusion) during the course of the study.
5. Subjects must be free of any systemic or dermatologic disorder, which in the opinion of the Investigator, will interfere with the study results.
6. Female subjects of childbearing potential must agree to use contraception during the study. All women of childbearing potential must have a negative urine pregnancy test at Screening and Baseline and at 4, 8 & 12 weeks visits.
7. Subjects are physically able to apply study product to all affected areas or can obtain help.

Exclusion Criteria:

1. Women who are pregnant or nursing or planning to become pregnant during the study.
2. Subjects who have been treated for warts within the 30 days prior to the Baseline Visit (e.g. salicylic acid, azelaic acid, cryotherapy).
3. Subjects who have participated in a trial involving any investigational product in the 30 days prior to the Baseline Visit.
4. Subjects with chronic or active liver disease, renal impairment, cutaneous or systemic lupus erythematosus, an autoimmune disorder, immunosuppression, or any other disease or medical condition that would interfere with the study or place the subject at unacceptable risk, as determined by the investigator.
5. Subjects on immunosuppressive agents that would impact their immune response e.g. cyclosporine, mycophenolate mofetil, azathioprine, etc.
6. Subjects who use or have used local/systemic steroids or any other immunosuppressive medication within the 30 days prior to the Baseline Visit.
7. Subjects who use or have used systemic or topical retinoids within the 30 days prior to the Baseline Visit.
8. Subjects who are unable to comply with study requirements.
9. Subjects with other skin diseases like molluscum contagiosum that may confound the evaluation of common warts.
10. Subjects who have received treatment for any type of cancer within 5 years of the Baseline Visit, except skin cancer and cervical cancer (in situ) are allowed if at least 1 year before the Baseline Visit.
11. Subjects unable to comply with study requirements

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects categorized as treatment responders (defined as having at least 91% reduction in surface area, averaged across all target warts) | Visit 5 (week 12)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Investigation Site #1, Hot Springs, Arkansas
  - Investigational Site #4, Fremont, California
  - Investigational Site #11, Sacramento, California
  - Investigational Site #2, Colorado Springs, Colorado
  - Investigational Site #12, Tampa, Florida
  - Investigational Site #9, Marietta, Georgia
  - Investigational Site #3, Arlington Hts, Illinois
  - Investigational Site #10, Crowley, Louisiana
  - Investigational Site #8, Fridley, Minnesota
  - Investigational Site #6, Johnston, Rhode Island
  - Investigational Site #5, Austin, Texas
  - Investigational Site #7, College Station, Texas